CLINICAL TRIAL: NCT01801878
Title: Pilot Study of Skin Quality Improvement After Adipose-drived Stem Cell Transfer in Irradiated Breasts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting research subjects
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B-1206-158-005; 06-2012-193 (Other: HurimBiocell, Inc)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Breast Neoplasms; Skin Abnormalities
Keywords: breast cancer; loss of elasticity in irradiated breast skin; Other Reconstructive Surgery
MeSH Terms: conditions — Breast Neoplasms; Skin Abnormalities | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose SVF cell (Experimental): adipose SVF cell transfer to the half of irradiated breast
  Interventions: Biological: Adipose SVF cell
- Normal saline (Active Comparator): Normal saline inject to the half of irradiated breast
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Adipose SVF cell — adipose SVF cell transfer to the half of irradiated breast
  Arms: Adipose SVF cell
Biological: Normal saline — Normal saline inject to the half of irradiated breast
  Arms: Normal saline

SUMMARY:
The aim of this study is to evaluate the skin quality of using adipose-drived stromal vascular fraction (SVF) cell taken by automatic centrifuge for adipose-drived cell isolation system into irradiated breasts.

DETAILED DESCRIPTION:
10 participants who taken conservative mastectomy will be enrolled

1. Process

   * adipose tissue is obtained from the subject's thigh or abdomen
   * adipose-drived stromal vascular fraction(SVF)cell isolation using automatic centrifuge system
   * adipose-drived stromal vascular fraction(SVF)cell graft into the irradiated breast.
2. Duration of study

   * entire duration: approximate 30weeks
   * Follow-up period: 12 weeks
   * Enrollment period: 12 weeks
3. Study design - Randomized, prospective, pilot study

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 40 and 60
* Subjects who diagnosed breast ductal carcinoma in situ of surgical staging T1aN0, negative resection margin of below 2mm in histopathologic examination
* Subjects who have a relapse-free interval of more than one year after breast-conserving surgery for breast cancer and radiation therapy
* Subjects who understand the study contents and sign the informed consent

Exclusion Criteria:

* Subjects who have radiodermatitis
* Subjects who planned breast reconstruction with autogenous tissue (ex.Transverse Rectus Abdominis Muscle flap)
* Subjects who have a history of smoking within 3months recently
* Subjects who participated in other clinical trial within 30 days recently
* Pregnant or lactating subjects
* Subjects who have a active infectious disease
* Subjects who are not eligible for this study at the discretion of the investigator

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The change in the breast skin thickness of the pre and post SVF graft from baseline at 12week after procedure | change in the breast skin thickness from baseline at 12 week
  The efficacy is assessed by breast skin thickness measured by radiologist using breast ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong Heo, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Bundang,Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided